CLINICAL TRIAL: NCT00995852
Title: Unilateral vs. Bilateral IBV Placement
Brief Title: Unilateral Versus Bilateral Endoscopic Lung Volume Reduction A Comparative Case Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Olympus Corporation of the Americas (Industry)
Responsible Party: Prof. Felix JF Herth, Thoraxklinik Heidelberg
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09 2009
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2009-10

CONDITIONS: Pulmonary Emphysema
Keywords: Endoscopic lung volume reduction; emphysema; COPD; Patients with bilateral heterogeneous pulmonary emphysema
MeSH Terms: conditions — Pulmonary Emphysema; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bilateral (Active Comparator): Treatment arm B - incomplete bilateral treatment of in total two lobes (contralateral).
  The study will only use Intrabronchial Valves™
  Interventions: Device: IBV Implantation
- unilateral (Active Comparator): Treatment arm A - unilateral treatment with complete closure of the worst lobe of the lungs
  Interventions: Device: IBV Implantation

INTERVENTIONS:
Device: IBV Implantation — In severe cases of COPD even optimum treatment involving bronchodilatation with drugs, physical training and possibly oxygen therapy is unable to influence exercise capacity and the perception of dyspnoea to a sufficient extent. Given the assumption that the elastic recoil of the small airways can be improved by a reduction in lung volume and pulmonary function overall by more ergonomic breathing mechanics and diaphragm function, various endoscopic procedures for lung volume reduction are available. Here one of the most advanced techniques is the implantation of intrabronchial valves. The one-way mechanism of this valve allows air to escape from the downstream lung segment without any influx of "new" air during inspiration
  Other Names: Spiration IBV
  Arms: unilateral
Device: IBV Implantation — In severe cases of COPD even optimum treatment involving bronchodilatation with drugs, physical training and possibly oxygen therapy is unable to influence exercise capacity and the perception of dyspnoea to a sufficient extent. Given the assumption that the elastic recoil of the small airways can be improved by a reduction in lung volume and pulmonary function overall by more ergonomic breathing mechanics and diaphragm function, various endoscopic procedures for lung volume reduction are available. Here one of the most advanced techniques is the implantation of intrabronchial valves. The one-way mechanism of this valve allows air to escape from the downstream lung segment without any influx of "new" air during inspiration
  Other Names: Spiration IBV
  Arms: bilateral

SUMMARY:
Patients with bilateral heterogeneous pulmonary emphysema benefit to differing degrees from unilateral ELVR with complete lobe closure in comparison with incomplete bilateral treatment.

DETAILED DESCRIPTION:
Patient enrolment and data acquisition is to be carried out on a prospective basis. It is planned to enrol a total of 20 patients with bilateral heterogeneous pulmonary emphysema. All patients will undergo treatment at one study centre in Heidelberg. Patients will be considered for both unilateral and bilateral treatment with intrabronchial valves (IBV) on the basis of their emphysema distribution. Patients will be randomised to two treatment arms. 10 patients receive unilateral or bilateral treatment in each case.

ELIGIBILITY:
Inclusion Criteria:

* age > 40 inhomogeneous emphysema FEV1 between 20-40% DLCO between 20-40% 6MWT > 150 m

Exclusion Criteria:

* pregnant homogeneous disease FEV1 < 20%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in pulmonary function (FEV1) 6-minute walking test | 3 months

SECONDARY OUTCOMES:
Number of major complications(SAE) | 3 months
Evaluation of the IBV migration rate | 3 months
Average changes in quality of life (SGRQ) | 3 months
Average changes in pulmonary function (FEV1, IVC, RV, TLC, RV/TLC) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Felix JF Herth, MD, Principal Investigator — Heidelberg University
Locations (1):
- Thoraxklinik Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Venuta F, Rendina EA, Coloni GF. Endobronchial treatment of emphysema with one-way valves. Thorac Surg Clin. 2009 May;19(2):255-60, x. doi: 10.1016/j.thorsurg.2009.04.002. PMID 19662969
- [Background] Chan KM, Martinez FJ, Chang AC. Nonmedical therapy for chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2009 Jan 15;6(1):137-45. doi: 10.1513/pats.200809-114GO. PMID 19131539
- [Background] Ingenito EP, Wood DE, Utz JP. Bronchoscopic lung volume reduction in severe emphysema. Proc Am Thorac Soc. 2008 May 1;5(4):454-60. doi: 10.1513/pats.200707-085ET. PMID 18453355
- [Derived] Eberhardt R, Gompelmann D, Schuhmann M, Reinhardt H, Ernst A, Heussel CP, Herth FJF. Complete unilateral vs partial bilateral endoscopic lung volume reduction in patients with bilateral lung emphysema. Chest. 2012 Oct;142(4):900-908. doi: 10.1378/chest.11-2886. PMID 22459779